CLINICAL TRIAL: NCT06479577
Title: Comparative Effects of Therapeutic Ultrasound and High Intensity Laser Therapy on Neuropathic Pain ,Strength and Quality of Life in Diabetic Foot
Brief Title: US & HILT Comparative Effect on Neuropathic Pain, Strength & QOF in Diabetic Foot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REC/RCR/23/02101 Zara Tariq
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Diabetic Foot; Diabetic Neuropathies
Keywords: diabetic neuropathies
MeSH Terms: conditions — Diabetic Foot; Diabetic Neuropathies | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound (Experimental): therapeutic ultrasound 1MHZ continuous mode for 20 minutes
  Interventions: Other: ultrasound
- high intensity laser therapy (Active Comparator): approximately 905 nm super pulsed laser
  Interventions: Other: high intensity laser therapy

INTERVENTIONS:
Other: ultrasound — ultrasound 1 MHZ continuous for 20 minute with routine physical therapy 3 days /week 150 minutes/ week resistance training 5-10 exercises involving major muscles of leg and foot 3-4 sets per exercise and 10- 15 repetition per set
  Arms: ultrasound
Other: high intensity laser therapy — 905 nm super pulsed laser 40 minute session 3 days /week 150 minutes/ week resistance training 5-10 exercises involving major muscles of leg and foot 3-4 sets per exercise and 10- 15 repetition per set
  Arms: high intensity laser therapy

SUMMARY:
To compare the effects of therapeutic ultrasound and high intensity laser therapy on neuropathic pain , strength and quality of life in patients with diabetic foot

DETAILED DESCRIPTION:
therapeutic ultrasound and laser therapy with routine physical therapy are used to improve neuropathic pain and foot related quality of life. the scarcity of evidence regarding the application of high intensity laser therapy necessitates a comprehensive investigation. The effects of HILT and comparative effects with ultrasound remains largely unexplored in diabetic peripheral neuropathy

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes.
* Diabetic Patients of age 50 to 75 years.
* Diabetic patient of Both genders
* Diagnosed Diabetes Mellitus with at least 7 years of duration
* Distal symmetrical or asymmetrical polyneuropathy with pain in the lower extremity for ≥6 months
* DNS (Diabetic neuropathy symptoms questionnaire) score greater than 4 (90 percent probability of neuropath

Exclusion Criteria:

* Pregnant females
* Lower limb Amputated patients
* History or evidence of neurological disorders other than peripheral neuropathy associated with Diabetes mellitus.

  * Evidence of musculoskeletal dysfunctions like scoliosis, lumbar disc prolapses and lumbar spine associated radiculopathy.
  * History of any low back surgeries and lower limb surgeries
* Patient with malignancy. Patient with epilepsy
* Patient with hemophilia
* Patient with pacemaker, metal implants prosthesis and internal fixation screws.
* Patient with severe cervical and lumbar neuropathy, rheumatoid arthritis, hereditary neuropathy
* Patient with a history of neurosurgery

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
michigan neuropathy screening instrument | 8th week
  MNSI is designed to screen for the presence of diabetic neuropathy the first part consist of 15 self administered questions on foot sensations ,pain ,numbness etc second part is brief physical examination of feet
foot and ankle disability index | 8th week
  FADI is designed to assess functional limitations related to foot and ankle conditions it has 26 items each item scored from 0 -4 FADI has totel 104 points

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, Phd, Principal Investigator — Riphah International University
Locations (1):
- Bahawalpur medical and dental hospital, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu Y, Xing P, Cai X, Luo D, Li R, Lloyd C, Sartorius N, Li M. Prevalence and Risk Factors for Diabetic Peripheral Neuropathy in Type 2 Diabetic Patients From 14 Countries: Estimates of the INTERPRET-DD Study. Front Public Health. 2020 Oct 20;8:534372. doi: 10.3389/fpubh.2020.534372. eCollection 2020. PMID 33194943
- [Background] Lin L, Li J, Lin J, Tang S, Li Y. Effectiveness and safety of low-level laser therapy in diabetic peripheral neuropathy: a protocol for a systematic review and meta-analysis. Syst Rev. 2021 Apr 2;10(1):96. doi: 10.1186/s13643-021-01656-y. PMID 33810813
- [Background] Tsiringakis G, Dimitriadis Z, Triantafylloy E, McLean S. Motor control training of deep neck flexors with pressure biofeedback improves pain and disability in patients with neck pain: A systematic review and meta-analysis. Musculoskelet Sci Pract. 2020 Dec;50:102220. doi: 10.1016/j.msksp.2020.102220. Epub 2020 Jul 24. PMID 32827852
- [Background] Eun IS, Oh YS, Kim J, Jang W. Reliability and Validity of the Korean Version of Foot and Ankle Disability Index. J Foot Ankle Surg. 2024 Jan-Feb;63(1):33-35. doi: 10.1053/j.jfas.2023.08.007. Epub 2023 Aug 19. PMID 37604317
- [Background] Seyedizadeh SH, Cheragh-Birjandi S, Hamedi Nia MR. The Effects of Combined Exercise Training (Resistance-Aerobic) on Serum Kinesin and Physical Function in Type 2 Diabetes Patients with Diabetic Peripheral Neuropathy (Randomized Controlled Trials). J Diabetes Res. 2020 Mar 6;2020:6978128. doi: 10.1155/2020/6978128. eCollection 2020. PMID 32215272